CLINICAL TRIAL: NCT03986970
Title: Combined HIV Adolescent PrEP and Prevention: On Demand Pre-exposure Prophylaxis to Provide Protection From HIV in Men - Using Foreskin Tissue to Estimate Protection (Phase II)
Brief Title: The CHAPS Trial: Combined HIV Adolescent PrEP and Prevention
Acronym: CHAPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wits Health Consortium (Pty) Ltd (Other)
Collaborators: University of Cape Town (Other); University of Liverpool (Other); Imperial College London (Other); MRC/UVRI Uganda Research Unit (Unknown); Karolinska Institutet (Other); King's College London (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: The CHAPS Trial
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2021-04

CONDITIONS: HIV/AIDS
Keywords: Pre-exposure prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Emtricitabine; tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Open-label, randomised controlled trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Arm 1: Control (No Intervention): No PrEP.
- Arm 2: FTC-TDF (Experimental): FTC-TDF one day, 5 hours before circumcision.
  Interventions: Drug: Tenofovir
- Arm 3: FTC-TDF (Experimental): FTC-TDF one day, 21 hours before circumcision.
  Interventions: Drug: Tenofovir
- Arm 4: FTC-TDF (Experimental): FTC-TDF two days, 5 hours before circumcision.
  Interventions: Drug: Tenofovir
- Arm 5: FTC-TDF (Experimental): FTC-TDF two days, 21 hours before circumcision.
  Interventions: Drug: Tenofovir
- Arm 6: FTC-TAF (Experimental): FTC-TAF one day, 5 hours before circumcision.
  Interventions: Drug: Tenofovir
- Arm 7: FTC-TAF (Experimental): FTC-TAF one day, 21 hours before circumcision.
  Interventions: Drug: Tenofovir
- Arm 8: FTC-TAF (Experimental): FTC-TAF two days, 5 hours before circumcision.
  Interventions: Drug: Tenofovir
- Arm 9: FTC-TAF (Experimental): FTC-TAF two days, 21 hours before circumcision.
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir — Pre-exposure prophylaxis
  Other Names: Emtricitabine, Tenofovir disoproxil, Tenofovir alafenamide
  Arms: Arm 2: FTC-TDF; Arm 3: FTC-TDF; Arm 4: FTC-TDF; Arm 5: FTC-TDF; Arm 6: FTC-TAF; Arm 7: FTC-TAF; Arm 8: FTC-TAF; Arm 9: FTC-TAF

SUMMARY:
To compare the effect of different PrEP drugs (FTC-TDF and FTC-TAF), doses and timing of doses on p24 antigen level in resected foreskin tissue following HIV exposure ex vivo challenge.

DETAILED DESCRIPTION:
1. Investigate the timing and dose of FTC-TDF and FTC-TAF as oral PrEP and in vitro PEP (applied directly to removed foreskin tissue) required to prevent ex vivo HIV infection in foreskin tissue and blood using the explant model
2. Determine blood, rectal fluid and foreskin tissue concentrations of FTC, TFV, TAF and their active metabolites that are required for ex vivo HIV protection
3. Evaluate inflammation, cellular activation, foreskin mucosal integrity, gene expression and microbiome in foreskin tissue following oral in vivo PrEP and in vitro PEP
4. Evaluate the efficacy of in vitro post exposure dosing with PrEP in protection against ex vivo HIV infection using the explant model
5. To investigate sexual behaviour, PrEP acceptability and feedback on HIV prevention trials implementation

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all the following criteria within 21 days prior to their circumcision visit:

1. Clinically eligible for either forceps guided, or dorsal slit circumcision
2. The ability to understand and sign a written informed consent form by participant (and participant's legal guardian if younger than 18 years) prior to participation in any study procedures and to comply with all trial requirements
3. Male sex at birth
4. Age 13- 24 years
5. Haemoglobin >9g/dL
6. Weight >35Kg
7. Two negative rapid HIV antibody tests results (manufactured by different companies), dating from 21 days or less prior to VMMC
8. Two locator information details (including physical address, telephone contacts, email) for contacting of either patient or their parent

Exclusion Criteria:

1. Any significant acute or chronic medical illness and current therapy that in the opinion of the site investigator would preclude receipt either of investigational products, or VMMC
2. Any evidence that participant is not suitable for VMMC

Ages: 13 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male genital anatomical features.
Enrollment: 72 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
HIV Infection free | 15 days
  We will ascertain the proportion of patients' foreskin tissue that is not infected with HIV 15 days following our ex-vivo HIV challenge. We will use the concentration of p24 antigen (pg/mL) at day15 and also report the slope of the p24 curves from day 3 to 15 (pg/mL per day) and also the AUC day 3 to 15 (pg/mL days).

SECONDARY OUTCOMES:
Timing | 1 year
  The delay between the timing of last dose of FTC-TDF and FTC-TAF as oral PrEP and the timing of circumcision.
Dose | 1 year
  The efficacy of preventing in-vitro HIV infection by dose of FTC-TDF and FTC-TAF as oral PrEP compared to no intervention
Blood PrEP Concentrations | 1 year
  Plasma concentrations (ng/mL) of FTC, TFV, TAF and their active metabolites that are required for ex vivo HIV protection.
Rectal Fluid PrEP concentrations | 1 year
  Rectal fluid concentrations (ng/mL) of FTC, TFV, TAF and their active metabolites that are required for ex vivo HIV protection.
Foreskin tissue PrEP concentration | 1 year
  Foreskin tissue concentrations (ng/mL) of FTC, TFV, TAF and their active metabolites that are required for ex vivo HIV protection
Efficacy of post-exposure PrEP | 1 year
  The proportion of participants' foreskin tissue that remains HIV infection free in the ex-vivo challenge model when additional doses of PrEP are added to that model.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Martinson, Principal Investigator — Perinatal HIV Research Unit
Locations (1):
- The Perinatal HIV Research Unit, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared with callaborators.

REFERENCES:
- [Derived] Nash S, Dietrich J, Ssemata AS, Herrera C, O'Hagan K, Else L, Chiodi F, Kelly C, Shattock R, Chirenje M, Lebina L, Khoo S, Bekker LG, Weiss HA, Gray C, Stranix-Chibanda L, Kaleebu P, Seeley J, Martinson N, Fox J; CHAPS team. Combined HIV Adolescent Prevention Study (CHAPS): comparison of HIV pre-exposure prophylaxis regimens for adolescents in sub-Saharan Africa-study protocol for a mixed-methods study including a randomised controlled trial. Trials. 2020 Oct 30;21(1):900. doi: 10.1186/s13063-020-04760-x. PMID 33121503
- See also: Related Info — http://trialsjournal.biomedcentral.com/track/pdf/10.1186/s13063-020-04760-x.pdf
- See also: Related Info — https://www.croiconference.org/abstract/pharmacokinetic-and-pharmacodynamic-study-of-tfv-and-taf-for-prep-in-foreskin-tissue/